CLINICAL TRIAL: NCT06157905
Title: Efficacy and Safety of Oral Tofacitinib in the Treatment of Alopecia Areata
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Hira Tariq, Principal Investigator, Services Institute of Medical Sciences, Pakistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB/2022/996/SIMS
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Extensive Alopecia Areata
Keywords: alopecia areata; Tofacitinib; Efficacy; Safety; Hair loss
MeSH Terms: conditions — Alopecia Areata; Alopecia | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients of Extensive alopecia areata (Experimental): Patients of either gender, age between 18-60 years, having extensive alopecia areata (SALT>24)
  Interventions: Drug: Oral Tofacitinib citrate

INTERVENTIONS:
Drug: Oral Tofacitinib citrate — oral tofacitinib citrate was initiated at 5 mg twice daily after ruling out contraindications

SUMMARY:
This clinical trial was conducted at the Dermatology department of Services hospital Lahore. Patients of extensive and treatment resistant Alopecia areata were enrolled after ethical approval and informed consent by non-probability consecutive sampling. Inclusion criteria: Treatment with oral tofacitinib citrate was initiated at 5 mg twice daily for six months. Scalp hair loss was calculated at 4, 12 and 24 weeks using the validated Severity of Alopecia Tool (SALT) score, which ranges from 0% to 100%. Regrowth rate: (initial SALT score - final SALT score)/(initial SALT score) × 100 was noted. Response time (time from initiation of treatment to any sign of hair regrowth) was noted. DLQI of patients before and after treatment were noted. Side effects were noted. Pre- and post-treatment photographs were taken. Patients were followed up for another 6 months to look for relapse.

Data were entered and analyzed using SPSS 20. Means were calculated for quantitative variables, frequencies for qualitative data. Data were stratified for the role of effect modifiers.

DETAILED DESCRIPTION:
This clinical trial was conducted at the Dermatology department of Services hospital Lahore. Patients of extensive and treatment resistant Alopecia areata were enrolled after ethical approval and informed consent by non-probability consecutive sampling. Treatment with oral tofacitinib citrate was initiated at 5 mg twice daily for six months after labs and ruling out contraindications. Scalp hair loss was calculated at 4, 12 and 24 weeks using the validated Severity of Alopecia Tool (SALT) score, which ranges from 0% to 100%. Regrowth rate: (initial SALT score - final SALT score)/(initial SALT score) × 100 was noted. Response time (time from initiation of treatment to any sign of hair regrowth) was noted. DLQI of patients before and after treatment were noted. Side effects were noted. Pre- and post-treatment photographs were taken. Patients were followed up for another 6 months to look for relapse.

Data were entered and analyzed using SPSS 20. Means were calculated for quantitative variables, frequencies for qualitative data. Data were stratified for the role of effect modifiers.

ELIGIBILITY:
Inclusion Criteria:

* Either gender Age 18 to 60 years Extensive disease (SALT > 24)

Exclusion Criteria:

* Patients taking immunosuppressants or DMARDs Recent live vaccination Active or latent TB, Hepatitis B or C, HIV Malignancy Hypersensitivity to the drug Pregnant or lactating mothers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2022-08-06 (Actual); Primary Completion 2023-02-05 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
50% reduction in Severity of Alopecia Tool (SALT) | within 24 weeks
  atleast 50% reduction of SALT score from baseline (pre-treatment)
50% reduction in Dermatology Life Quality Index (DLQI) | within 24 weeks
  Atleast 50% improvement in quality of life of patients by reduction in DLQI from baseline (pre-treatment)

OTHER OUTCOMES:
Regrowth rate | within 24 weeks
  (initial SALT score - final SALT score)/(initial SALT score) × 100
Response time | within 24 weeks
  time from initiation of treatment to any sign of hair regrowth

CONTACTS AND LOCATIONS:
Locations (1):
- Services Institute of Medical Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xing L, Dai Z, Jabbari A, Cerise JE, Higgins CA, Gong W, de Jong A, Harel S, DeStefano GM, Rothman L, Singh P, Petukhova L, Mackay-Wiggan J, Christiano AM, Clynes R. Alopecia areata is driven by cytotoxic T lymphocytes and is reversed by JAK inhibition. Nat Med. 2014 Sep;20(9):1043-9. doi: 10.1038/nm.3645. Epub 2014 Aug 17. PMID 25129481
- [Background] Jabbari A, Nguyen N, Cerise JE, Ulerio G, de Jong A, Clynes R, Christiano AM, Mackay-Wiggan J. Treatment of an alopecia areata patient with tofacitinib results in regrowth of hair and changes in serum and skin biomarkers. Exp Dermatol. 2016 Aug;25(8):642-3. doi: 10.1111/exd.13060. No abstract available. PMID 27119625